CLINICAL TRIAL: NCT05427474
Title: Role of Combined Therapy of Propranolol and Gabapentin in Paroxysmal Sympathetic Hyperactivity in Traumatic Brain Injury at Emergency Intensive Care Unit
Brief Title: Role of Combined Therapy of Propranolol and Gabapentin in Paroxysmal Sympathetic Hyperactivity in Traumatic Brain Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Essamedin Mamdouh Negm, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9076-8-11-2021
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol; Gabapentin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard protocol of manaegement (No Intervention): traumatic brain injury protocol in Emergency ICU without adding propranolol or gabapentin
- propranolol group (Active Comparator): addding propranolol to the traumatic brain injury protocol in Emergency ICU
  Interventions: Drug: Propranolol , gabapentin
- combined propranolol and gabapentin (Active Comparator): adding propranolol and gabapentin to the traumatic brain injury protocol in Emergency ICU
  Interventions: Drug: Propranolol , gabapentin

INTERVENTIONS:
Drug: Propranolol , gabapentin — The combined therapy of propranolol and gabapentine can prevent the occurrence of paroxysmal sympathetic hyperactivity in traumatic brain injury patients and improve the clinical outcomes in emergency ICU.
  Arms: combined propranolol and gabapentin; propranolol group

SUMMARY:
Paroxysmal sympathetic hyperactivity (PSH) is a syndrome that comprises a series of signs and symptoms reflecting exacerbated sympathetic activity, including arterial hypertension, fever, tachycardia, generalized perspiration, anomalous motor activity (dystonia, muscle stiffness, extension), tachypnea, mechanical ventilator maladjustment, hypoxemia, hypercapnia, and hyperglycemia. PSH episodes can be intense and prolonged and can occur several times a day and all of these can lead to secondary brain damage and are the main causes of a poor prognosis. Paroxysmal sympathetic hyperactivity also induces a hypermetabolic state with hypercatabolism and inflammation and increases vulnerability to infections, sepsis, and weight loss which in turn are associated with increased morbidity, longer hospital stay, and slower recovery. The marked and sustained increase in catecholamine levels predisposes to the development of cardiomyopathy, lung edema, arrhythmias, and cardiac and multisystemic dysfunction.

The reported incidence of paroxysmal sympathetic hyperactivity ranges from 8% to 33% and has no particular age or gender predilection. 80% of these syndrome incidents developed with traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a critical public health problem worldwide. It has been referred to as the " silent epidemic " as the problems experienced by those patients (such as impairments in memory or cognition) are often not visible.

According to the World Health Organization, traumatic brain injury will surpass many diseases as the major cause of death and disability. Each year an estimated 69 million individuals will suffer a TBI, the vast majority of which will be mild (81%) and moderate (11%) in severity. Many survivors live with significant disabilities, resulting in a major socioeconomic burden.

Nearly 60% of traumatic brain injuries are due to road traffic injuries in all parts of the world, about 20-30% are due to falls, 10% due to violence, and another 10% due to a combination of workplace and sports-related injuries.

Paroxysmal sympathetic hyperactivity (PSH) is a syndrome that comprises a series of signs and symptoms reflecting exacerbated sympathetic activity, including arterial hypertension, fever, tachycardia, generalized perspiration, anomalous motor activity (dystonia , muscle stiffness, extension), tachypnea, mechanical ventilator maladjustment, hypoxemia, hypercapnia, and hyperglycemia (Hughes and Rabinstein,2014). PSH episodes can be intense and prolonged and can occur several times a day and all of these can lead to secondary brain damage and are the main causes of a poor prognosis. Paroxysmal sympathetic hyperactivity also induces a hypermetabolic state with hypercatabolism and inflammation and increases vulnerability to infections, sepsis, and weight loss which in turn are associated with increased morbidity, longer hospital stay, and slower recovery. The marked and sustained increase in catecholamine levels predisposes to the development of cardiomyopathy, lung edema, arrhythmias, and cardiac and multisystemic dysfunction.

The reported incidence of paroxysmal sympathetic hyperactivity ranges from 8% to 33% and has no particular age or gender predilection. 80% of these syndrome incidents developed with traumatic brain injury.

Paroxysmal sympathetic hyperactivity manifests suddenly in cyclic episodes either spontaneously or in response to stimuli like pain, bathing, suction of secretions, exposure to light, and touch.

Paroxysmal sympathetic hyperactivity is a genuine neurological emergency that may go undetected if not taken into account. An early diagnosis and optimized treatment are crucial in order to avoid permanent disability, reduce complications rate, facilitate recovery, and shorten stay in the intensive care unit.

Because of the complexity of the disease and as its etiology is not clearly understood so pharmacological therapy has focused on the control of symptoms.

It is important to note the lack of studies demonstrating the preference of one drug substance versus another. The experience and the literature indicate that "drug combinations" are generally required.

Propranolol is a non-selective beta-blocker that can cross the blood-brain barrier; so many studies showed that early administration of propranolol after TBI was associated with improved survival, and also a large cohort study reported the benefit of propranolol as the preferred beta-blocker agent to be used to decrease the incidence of secondary brain injury and to improve mortality outcome in patients with TBI experiencing PSH.

Gabapentine, an analog of GABA was originally developed as an anticonvulsant. However, it may be more useful in the management of painful neuropathies, spasticity, and tremor. Administration of gabapentin before the neuropathic pain establishment showed a long-lasting anti-allodynic effect.

Studies show its dramatic effect on the improvement of the frequency and severity of the paroxysmal sympathetic hyperactivity spells within days of starting gabapentin which has become the first choice for the longer-term control of this disorder.

Rationale:

Paroxysmal sympathetic hyperactivity occurs after any brain lesion and has been associated with worse clinical outcomes including more time on mechanical ventilation, more infection, tracheostomy placement, longer ICU stay, and so increase mortality rate.

Medical treatments for PSH include Opioids like morphine, and fentanyl, Beta-blockers as propranolol, Alpha 2 agonists like dexmedetomidine, and GABA agonists as gabapentin and benzodiazepines and baclofen, and muscle relaxant dantrolene. This pharmacological management focuses on three approaches: symptom abortion, prevention of symptoms, and refractory treatment.

Up to the investigators' knowledge, this is the first study in zagazig university hospital to evaluate the success of the combined therapy of propranolol and gabapentin in preventing the development of PSH in traumatic brain injury patients.

Research question:

Can the combined therapy of propranolol and gabapentin prevent the occurrence of paroxysmal sympathetic hyperactivity and improve the clinical outcomes of traumatic brain injury patients in emergency ICU?

ELIGIBILITY:
Inclusion Criteria:

* • ICU patients with moderate (GCS 9-12) to severe (GCS <9) traumatic brain injury .

Exclusion Criteria:

* Pre-existing brain dysfunction .
* History of allergy to any of the combined drug therapy ( propranolol or gabapentine ) .
* History of obstructive lung disease .
* History of heart disease .
* Hypotension at admission of ICU.
* Bradycardia .
* Hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
mortality rate of patients | 8 months
  to record the mortality rate of each group of patients

SECONDARY OUTCOMES:
incidence of PSH | 8 months
  to calculate the incidence of paroxysmal sympathetic hyperactivity among moderate and severe traumatic brain injury patients who receive the combined therapy of propranolol and gabapentine in emergency ICU
ICU length of stay | 8 months
  to calculate the length of stay of patients for each group
conscious level | 8 months
  to determine GCS for patients for each group

CONTACTS AND LOCATIONS:
Overall Officials: Essamedin Negm, MD, Principal Investigator — Zagazig University
Locations (2):
- Egypt (2):
  - Zagazig University Hospitals, Zagazig
  - Zagazig University, Zagazig